CLINICAL TRIAL: NCT03188497
Title: Dose Escalation of Lobaplatin Concurrent With Intensity-modulated Radiotherapy for the Treatment of Stage III-IVb Nasopharyngeal Carcinoma: A Phase I Clinical Trial in an Asian Population
Brief Title: Dose Escalation of Lobaplatin Concurrent With IMRT for the Treatment of NPC: A Phase I Clinical Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fifth Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Xiwei XU, Clinical doctor, Fifth Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: zsu20170203
Record Dates: First submitted 2017-05-22; First posted 2017-06-15 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-04

CONDITIONS: Acute Toxic Effects; Tumor Responses
MeSH Terms: interventions — lobaplatin; Particle Accelerators

STUDY DESIGN:
Intervention Model Description: The initial dose was 25mg/m2 on d1,d22,d43 for 1 cycles; if no obvious toxicity was observed,follow 30mg/m2,35mg/m2,40mg/m2,45mg/m2, and 50mg/m2 gradients into the next dose group until the maximum tolerated dose or 50mg/m2
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experience group 1 (Experimental): The dose of lobaplatin is 25mg/m2 on d1,d22,d43.
  Interventions: Drug: Lobaplatin; Device: linear accelerator
- Experience group 2 (Experimental): The dose of lobaplatin is on d1,d22,d43.
  Interventions: Drug: Lobaplatin; Device: linear accelerator
- Experience group 3 (Experimental): The dose of lobaplatin is on d1,d22,d43.
  Interventions: Drug: Lobaplatin; Device: linear accelerator
- Experience group 4 (Experimental): The dose of lobaplatin is 40mg/m2 on d1,d22,d43.
  Interventions: Drug: Lobaplatin; Device: linear accelerator
- Experience group 5 (Experimental): The dose of lobaplatin is 45mg/m2 on d1,d22,d43.
  Interventions: Drug: Lobaplatin; Device: linear accelerator
- Experience group 6 (Experimental): The dose of lobaplatin is 50mg/m2 on d1,d22,d43.
  Interventions: Drug: Lobaplatin; Device: linear accelerator

INTERVENTIONS:
Drug: Lobaplatin — Lobaplatin for Injection
Device: linear accelerator — Medical linear accelerator

SUMMARY:
Nasopharyngeal carcinoma (NPC) is a common malignant tumor in Southern China area, which is characterized by obvious regional characteristics and "Guangdong cancer". Radiotherapy is the main treatment for locally advanced nasopharyngeal carcinoma. In recent years, chemotherapy has improved the short-term and long-term survival of patients with locally advanced nasopharyngeal carcinoma.

Lobaplatin is the third generation platinum anticancer drugs, mechanism of action and traditional cisplatin is similar, mainly formed by the Pt-GG and Pt-AG chain cross connect, replication and transcription process blocks of deoxyribonucleic acid(DNA), thereby interfering with tumor cell cycle. The damage of DNA induced by lobaplatin can influence the expression of tumor cell specific genes. Due to the different structure of lobaplatin and no cross resistance to cisplatin in the study showed that, compared with cisplatin with gastrointestinal reaction more mild, and no cisplatin common liver and kidney toxicity, neurotoxicity and ototoxicity, in some tumors have a better adaptability; but compared with cisplatin had more severe bone marrow suppression this, offset some of the advantages of lobaplatin in a certain extent. At present, the clinical indications for the treatment of such diseases include head and neck cancer, breast cancer, gastrointestinal cancer, gynecologic malignant tumor and non small cell lung cancer. Tian Ying confirmed that lobaplatin has obvious cytotoxic effect on nasopharyngeal carcinoma cells, in a concentration dependent manner, the mechanism for the dual role, namely block at lower concentration of cells in G2 phase and induce apoptosis at higher concentration, provide the possibility for clinical treatment of nasopharyngeal carcinoma for lobaplatin; there are a number of clinical study confirmed that lobaplatin chemoradiotherapy for locally advanced nasopharyngeal carcinoma with cisplatin approximation. But at present, there is no report on the dose and tolerability of concurrent radiotherapy for nasopharyngeal carcinoma.

Therefore, a dose escalation trial was conducted to determine maximum tolerated dose of lobaplat in as a single agent combined with concurrent intensity-modulated radiotherapy in a Chinese population with locoregionally advanced NPC.

ELIGIBILITY:
Inclusion Criteria:

1. The pathological type is non keratinized carcinoma (according to the pathological classification of World, Health, Organization, WHO)
2. Overall Stage III-IVB (according to the seventh edition of AJCC staging system).
3. Age between 18-65 years old.
4. There is no evidence of distant metastasis.
5. Eastern Cooperative Oncology Group performance status 0 or 1.
6. Normal marrow function: white blood count > 4 * 109/L, hemoglobin > 90g/L, and platelet count > 100 * 109/L.
7. Normal liver function: total bilirubin (TBIL) and alanine aminotransferase (ALT) <2 times the normal values.
8. Normal renal function: creatinine (Cr) <1.5 times the normal value.
9. The patient must be the basic content of this research and the defendant signed the informed consent.

Exclusion Criteria:

1. The pathological type is WHO squamous cell carcinoma or squamous cell carcinoma.
2. Age > 65 years old, or < 18 yeas old.
3. The purpose of treatment is palliative.
4. There was a history of malignancy, except for adequately treated basal cell carcinoma or squamous cell carcinoma, and carcinoma in situ of the cervix.
5. Women who are pregnant or lactating (for women of child-bearing age) should consider pregnancy tests; effective contraception should be emphasized during treatment）.
6. Previously received radiation therapy .
7. Primary and neck metastases were treated with chemotherapy or surgery.
8. Accompanied by other serious diseases may pose a greater risk or impact on test compliance.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-06-22 (Actual); Primary Completion 2017-12-12 (Actual); Study Completion 2018-03-20 (Actual)

PRIMARY OUTCOMES:
Platelets | 1 years
  grade 3: 25.0-< 50.0*109/L; grade 4:< 25.0*109/L.
Leukocytes | 1 years
  grade 3: 1.0-< 2.0*10^9/L; grade 4: < 1.0*10^9/L.
Neutrophils | 1 years
  grade 3: 0.5-< 1.0*10^9/L; grade 4: < 0.5*10^9/L.
Hemoglobin | 1 years
  grade 3: < 80 g/L; transfusion indicated; grade 4:Life-threatening consequences; urgent intervention indicated; grade 5: Death

SECONDARY OUTCOMES:
Nausea | 1 years
  grade 3: Inadequate oral caloric or fluid intake; tube feeding, TPN, or hospitalization indicated
Vomiting | 1 years
  grade 3: > 6 episodes (separated by 5 minutes) in 24 hrs; tube feeding, TPN, or hospitalization indicated; grade 4:Life-threatening consequences; urgent intervention indicated; grade 5: Death.

OTHER OUTCOMES:
Aspartate transaminase (ALT) | 1 years
  ALT: grade 3: > 5.0-20.0*ULN; grade 4: > 20.0*ULN.
Aspartate transaminase (AST) | 1 years
  grade 3: > 5.0-20.0*ULN; grade 4: > 20.0*ULN.
Bilirubin | 1 years
  grade 3: > 3.0-10.0*ULN; grade 4: > 10.0*ULN.
Glutamyl transpeptidase (GGT) | 1 years
  grade 3: > 5.0-20.0*ULN; grade 4: > 20.0*ULN.
Alkaline phosphatase (ALP) | 1 years
  grade 3:> 5.0-20.0*ULN; grade 4: > 20.0*ULN.
Creatinine（CRE） | 1 years
  grade 3: > 3.0-6.0*ULN, > 3.0 baseline; grade 4: > 6.0*ULN.

CONTACTS AND LOCATIONS:
Overall Officials: Siyang Wang, bachelor, Study Director — Fifth Hospital Affiliated to Sun Yet Sen universty
Locations (1):
- the Fifth Hospital Affiliated to Sun Yat-Sen University, Zhuhai, Guangdong, China

REFERENCES:
- [Derived] Wang SY, Xu XW, Yao JJ, Peng PJ, Zhou B, Liu QD, Huang XP, Lin Z. Dose Escalation of Lobaplatin Concurrent with IMRT for the Treatment of Stage III-IVb NPC: A Phase I Clinical Trial. Transl Oncol. 2018 Aug;11(4):1007-1011. doi: 10.1016/j.tranon.2018.06.004. Epub 2018 Jun 29. PMID 29966863